CLINICAL TRIAL: NCT07223606
Title: Fecal Microbiota Transplant for Neuroblastoma in a Single Patient
Status: No longer available | Type: Expanded Access
Sponsor: ProgenaBiome (Other)
Collaborators: Microbiome Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IND 31935; IND 31935 (Other: FDA)
Record Dates: First submitted 2025-09-18; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-09

CONDITIONS: Neuroblastoma; Neuroblastoma (NB); Neuroblastoma (NBL); Neuroblastoma (Measurable Disease); Neuroblastoma Recurrent; Neuroblastoma in Children; Neuroblastoma. CNS
Keywords: FMT; fecal transplant; fecal microbiota transplant; microbiome; dysbiosis
MeSH Terms: conditions — Neuroblastoma; Dysbiosis

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Fecal Microbial Transplantation — This study will utilize donor stool from an infant
  Other Names: FMT

SUMMARY:
This study uses fecal microbiota transplant (FMT) to correct gut microbiome dysbiosis prior to and during standard-of-care neuroblastoma treatment

DETAILED DESCRIPTION:
Patients with neurobastoma and concurrent dysbiosis showing a bifidobacteria-bacteroides gap will undergo fecal microbiota transplant as an adjunctive to standard-of-care oncology treatment.

ELIGIBILITY:
Inclusion Criteria:

* willingness of parent/guardian to sign ICF
* diagnosis of neuroblastoma
* dysbiosis of the gut microbiome

Exclusion Criteria:

* parent/guardian unwilling to sign ICF
* dysbiosis does not show a bifidobaceteria-bacteroides gap
* severely abnormal screening lab values

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- ProgenaBiome, Ventura, California, United States